CLINICAL TRIAL: NCT06721689
Title: A Phase 1/2 Clinical Trial of the Novel Topoisomerase I Inhibitor PEEL-224 as a Single Agent and in Combination With Vincristine and Temozolomide in Children With Refractory, Progressive or Relapsed Solid Tumors
Brief Title: PEEL-224, Vincristine and Temozolomide in Pediatric Solid Tumors
Acronym: PEEL-224
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theodore Laetsch (Other)
Collaborators: Peel Therapeutics Inc (Industry)
Responsible Party: Sponsor-Investigator, Theodore Laetsch, Director, Developmental Therapeutics Program and Very Rare Malignant Tumors Program, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-022741
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Refractory Solid Tumors; Relapsed Solid Tumors; Relapsed Neuroblastoma; Refractory Neuroblastoma; Relapsed Rhabdomyosarcoma; Refractory Rhabdomyosarcoma
Keywords: Relapsed; Refractory; Solid Tumor
MeSH Terms: conditions — Neuroblastoma; Rhabdomyosarcoma; Recurrence | interventions — Vincristine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEEL-224 (Experimental): Phase 1A will test the safety, tolerability and PK profile of PEEL-224 as a single agent in pediatric patients with refractory, progressive and relapsed solid tumors.
  Interventions: Drug: PEEL-224
- PEEL-224, Vincristine, and Temozolomide (Experimental): Phase 1B will test the safety, tolerability and pharmacokinetic profile of PEEL-224 in combination with vincristine and temozolomide in pediatric subjects with refractory, progressive and relapsed solid tumors. Phase 2 will preliminary evaluate the activity profile of PEEL-224 in combination with vincristine and temozolomide in pediatric patients with refractory, progressive and relapsed NBL and RMS.
  Interventions: Drug: PEEL-224; Drug: Vincristine; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: PEEL-224 — PEEL-224 (PEG-[SN22]4) is a novel topoisomerase I inhibitor
Drug: Vincristine — Vincristine is an inhibitor of microtubular formation which is approved by the Food and Drug Administration (FDA) and is commercially available.
  Arms: PEEL-224, Vincristine, and Temozolomide
Drug: Temozolomide (TMZ) — Temozolomide is an alkylating agent which is approved by the FDA and is commercially available.
  Arms: PEEL-224, Vincristine, and Temozolomide

SUMMARY:
The phase 1 primary objective is to determine the pediatric recommended phase 2 dose (RP2D) of PEEL-224 as a single agent (phase 1A) and in combination with vincristine and temozolomide (phase 1B). The phase 2 primary objective is to estimate the objective response rate (ORR) in children with refractory, progressive and relapsed NBL and rhabdomyosarcoma (RMS) treated with the RP2D of PEEL-224 in combination with vincristine and temozolomide.

DETAILED DESCRIPTION:
PEEL-224 will be a multi-institutional study conducted at pediatric cancer centers. Phase 1 will enroll approximately 24 subjects (maximum of 12 evaluable subjects in phase 1A and 12 evaluable subjects in phase 1B) between ages 1 to 18 years of age with a refractory, progressive or relapsed solid tumor. Phase 2 will enroll a maximum of 18 evaluable subjects with refractory, progressive or relapsed NBL and a maximum of 17 evaluable subjects with refractory, progressive or relapsed RMS. PEEL-224 will be administered at the assigned dose on days 1 and 8 of 21-day cycles as a single agent (phase 1A) or in combination with vincristine on days 1 and 8 and temozolomide on days 1-5 (phase 1B and phase 2). Subjects may continue protocol therapy for up to 24 cycles (approximately 18 months) in the absence of progressive disease or unacceptable toxicity. Subjects will be monitored with physical exams and labs on days 1 and 8 of each cycle and disease response assessments and patient reported outcome assessments will be performed after cycles 2, 4, 6, 9, 12, 18, and 24. During phase 1, PK blood samples will be drawn during cycle 1. The primary phase 1 endpoints are cycle 1 dose limiting toxicity (DLT) to define the RP2D. The primary phase 2 endpoint is best overall objective response to define the ORR.

ELIGIBILITY:
Inclusion Criteria:

1. Age:

   * Phase 1: Age greater than or equal to 1 year and less than or equal to18 years
   * Phase 2 Neuroblastoma (NBL) cohort: Age greater than or equal to 1 year and less than or equal to 30 years
   * Phase 2 Rhabdomyosarcoma (RMS) cohort: Age greater than or equal to 1 year and less than or equal to18 years
2. Diagnosis of:

   * Phase 1: Refractory, progressive or relapsed non-central nervous system (CNS) solid tumors who have received at least 1 line of upfront therapy. Patients must have had histologic verification of their malignancy at original diagnosis or relapse
   * Phase 2: Refractory, progressive or relapsed neuroblastoma (NBL) or rhabdomyosarcoma (RMS) who have received at least 1 line of upfront therapy. Patients must have had histologic verification of their malignancy at original diagnosis or relapse.
3. Disease status:

   * Phase 1: evaluable or measurable disease
   * Phase 2, subjects with Neuroblastoma (NBL): evaluable or measurable disease by International Neuroblastoma Response Criteria (INRC); subjects with only bone marrow disease are not eligible
   * Phase 2, subjects with rhabdomyosarcoma (RMS): measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST)1.1.
4. Adequate available archival tumor tissue as described in Section 5.4.3. Tumor tissue from the most recent biopsy or resection is preferred, if adequate sample is available. If no archival tumor tissue is available, enrollment may be permitted with prior approval by the overall study PI or designee.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 (age greater than 16 years) or Lansky Performance Status of at least 60 (age less than 16 years).
6. Females of childbearing potential must have a negative urine/serum pregnancy test.
7. Adequate bone marrow function

   Hematologic requirements for all subjects on phase 1 and subjects on phase 2 without malignant infiltration of the bone marrow:
   * Absolute neutrophil count (ANC) greater than or equal to 750/mm3 (greater than or equal to 7 days since last dose of short acting myeloid growth factor medications (e.g. filgrastim) and greater than or equal to 14 days since last dose of long-acting myeloid medications (e.g. peg-filgrastim)
   * Platelet count ≥ 75,000 mm3 (greater than or equal to 14 days since last dose of thrombopoietin receptor agonist such as romiplostim and without platelet transfusion within previous 7 days)
   * Not refractory to packed red blood cell transfusions

   Hematologic requirements for subjects on phase 2 with malignant infiltration of the bone marrow:
   * Absolute neutrophil count (ANC) greater than or equal to 500/mm3 (greater than or equal to 7 days since last dose of short acting myeloid growth factor medications (e.g. filgrastim) and greater than or equal to 14 days since last dose of long-acting myeloid medications (e.g. peg-filgrastim))
   * Platelet count greater than or equal to 50,000/mm3 (greater than or equal to 14 days since last dose of thrombopoietin receptor agonist such as romiplostim and without platelet transfusion within previous 7 days)
   * Not refractory to packed red blood cell transfusions
   * Patients on phase 2 with malignant infiltration of the bone marrow will not be evaluable for hematologic toxicity.
8. Adequate renal function as evidenced by creatinine clearance as calculated by the Schwartz equation (see below), radioisotope glomerular filtration rate (GFR) greater than or equal to 70 mL/min/1.73 m2, or maximum serum creatinine as below:

   Age Maximum Serum Creatinine (mg/dL)

   Male Female 1 to less than 2 years 0.6 0.6 2 to less than 6 years 0.8 0.8 6 to less than 10 years 1 1 10 to less than 13 years 1.2 1.2 13 to less than 16 years 1.5 1.4 greater than 16 years 1.7 1.4 Threshold derived from the Schwartz formula for estimating glomerular filtration rate (GFR) (Schwartz et al., J.Peds, 106:522,1985) utilizing child length and stature data published by the CDC The Schwartz equation for subjects less than 18 years of age: eGFR (mL/min/1.73 m2) = 0.413 x [height (cm)/serum creatinine (mg/dL)]
9. Adequate liver function

   * Aspartate Aminotransferase (AST/SGOT): less than or equal to 3 times the upper limit of normal (ULN) or less than or equal to 5 the upper limit of normal if attributable to disease involvement. For the purpose of this study, the upper limit of normal (ULN) for Aspartate Aminotransferase (AST) is 50 U/L.
   * Alanine Aminotransferase (ALT/SGPT): less than or equal to 3 times the ULN or less than or equal to 5 the upper limit of normal if attributable to disease involvement. For the purpose of this study, the upper limit of normal (ULN) for Alanine Aminotransferase (ALT) is 45 U/L.
   * Total bilirubin: less than or equal to 1.5 times the upper limit of normal with the exception of patients with Gilbert's syndrome who must have bilirubin less than 3X institutional upper limit of normal (ULN).
10. Prior Therapy: Patients must have had resolution of acute toxic effects of prior therapy to grade less than or equal to 1 according to the National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) v 5.0 except organ function as noted above, adverse events (AE) that are considered clinically non-significant (i.e. alopecia), or controlled on supportive care (i.e. nausea/vomiting, hypothyroidism). Patients must meet the following minimum washout periods prior to enrollment:

    * Myelosuppressive chemotherapy: At least 14 days after the last dose of myelosuppressive chemotherapy
    * Small molecule targeted therapy: At least 7 days following the last dose of a small molecule targeted agent.
    * Antibody therapy: At least 21 days following the last dose of antibody including anti-GD2 monoclonal antibody.
    * Cellular therapy: At least 42 days following completion of a cellular therapy agent (e.g. modified T cells, NK cells, dendritic cells)
    * Autologous hematopoietic stem cell transplant and stem cell boost: Subjects must be at least 60 days from day 0 of an autologous stem cell transplant or stem cell boost.
    * Myeloid growth factors: At least 7 days following short-acting myeloid growth factor (e.g. filgrastim) and at least 14 days following the last dose of long-acting myeloid growth factor (e.g. peg-filgrastim)
    * Thrombopoietin receptor agonists: At least 14 days following last dose of thrombopoietin receptor agonist such as romiplostim
    * Interleukins, interferons, and cytokines (other than hematopoietic growth factors): At least 21 days following the completion of interleukins, interferon, or cytokines, including IL-2
    * Radiotherapy:

      * At least 14 days after limited field radiation therapy;
      * At least 90 days after total body irradiation, craniospinal radiotherapy; or radiation to greater than 50% of pelvis;
      * At least 42 days must have elapsed if other substantial BM radiation.
    * Radiopharmaceutical therapy (e.g. radiolabeled antibody, 131I- MIBG): At least 42 days after radiopharmaceutical therapy
    * Major Surgery: At least 2 weeks from prior major surgical procedure. Note: Biopsy, CNS shunt placement/revision, and central line placement/removal are not considered major.
    * Strong CYP1A2 and/or CYP3A4 inhibitors and/or inducers: At least 14 days following use of a strong CYP1A2 and/or CYP3A4 inhibitor and/or inducer. See Appendix 1 for examples. (Note that levofloxacin is permitted when clinically indicated)
11. Prior treatment with irinotecan and/or temozolomide is permitted.
12. Female patients of reproductive potential must agree to use a highly effective contraceptive method for the duration of study therapy and for at least six months after the final dose of PEEL-224. Males of reproductive potential with a female partner of child-bearing potential must use a highly effective for the duration of the study and for at least six months after the final dose of PEEL-224.
13. Subjects must agree to use sun protective measures while receiving treatment and for 4 weeks after the last dose of PEEL-224
14. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Prior treatment with PEEL-224.
2. Subjects receiving any other anti-cancer agents.
3. Subjects with primary central nervous system (CNS) solid tumors or central nervous system (CNS) metastatic disease.
4. Subjects with prior allogeneic stem cell or solid organ transplantation.
5. Pregnant or lactating females.
6. Subjects with a known history of human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C (testing not required as part of screening).
7. Subjects with symptomatic congestive heart failure.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-03-23 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Phase 1A and Phase 1B: Number of participants who experience a dose limiting toxicity (DLT) | 1 month
  The observation of a dose-limiting toxicity (DLT) or lack of observation of DLT in the period between treatment initiation up to initiation of cycle 2 treatment. A dose limiting toxicity (DLT) describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Phase 2 Neuroblastoma Cohort (NBL): Number of paricptants who achieve a complete response (CR), partial response (PR), or minor response (MR) | 2 years
  Objective response as assessed by the Revised International Neuroblastoma Response Criteria (INRC). Response is defined as complete response (CR), partial response (PR) or minor response (MR), using best response measured at any point prior to local control.
Phase 2 Rhabdomyosarcoma (RMS) Cohort: Number of participants who achieve a complete response (CR) or partial response (PR) | 2 years
  Objective response as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. Response is defined as complete response (CR) or partial response (PR), using best response measured at any point prior to local control.

SECONDARY OUTCOMES:
Number of subjects with an Adverse Event (AE) of greater than or equal to grade 3 at least possibly attributable to study treatment | 30 days after last dose
  Adverse Events (AEs) will be graded by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Area under the plasma-concentration-time-curve of PEEL-224 | 1 month
  To characterize the pharmacokinetic (PK) profile of free SN22 and SN22 bound to PEG (PEEL-224)
Number of participants demonstrating anti-tumor activity of PEEL-224 | 2 years
  To preliminarily evaluate antitumor activity of PEEL-224 by estimating event-free survival (EFS)
Number of participants demonstrating anti-tumor activity of the combination of PEEL-224, vincristine and temozolomide | 2 years
  To preliminarily evaluate antitumor activity of the combination of PEEL-224, vincristine and temozolomide by estimating event-free survival (EFS )

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn Crane, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No